CLINICAL TRIAL: NCT02186951
Title: Prevention of Early Ventilator-associated Pneumonia With Antibiotic Therapy in Patients Treated With Mild Therapeutic Hypothermia After Cardiac Arrest.
Brief Title: Antibiotherapy During Therapeutic Hypothermia to Prevent Infectious Complications
Acronym: ANTHARTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I13018 ANTHARTIC
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Ventilator-associated Pneumonia; Cardiac Arrests With Shockable Rhythm; Mild Therapeutic Hypothermia; Preventive Antibiotics
Keywords: ventilator-associated pneumonia; cardiac arrests with shockable rhythm; Mild therapeutic hypothermia; preventive antibiotics
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin clavulanic acid (Experimental): Amoxicillin-clavulanic acid 1g, three times a day during 2 days, started within one hour after randomization and before the beginning of hypothermia.
  Interventions: Drug: Amoxicillin - clavulanic acid
- Placebo (Placebo Comparator): Placebo 1g, three times a day during 2 days, started within one hour after randomization and before the beginning of hypothermia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin - clavulanic acid — Amoxicillin-clavulanic acid 1g, three times a day during 2 days, started within one hour after randomization and before the beginning of hypothermia.
  Arms: Amoxicillin clavulanic acid
Drug: Placebo — Placebo 1g, three times a day during 2 days, started within one hour after randomization and before the beginning of hypothermia.
  Arms: Placebo

SUMMARY:
Mild therapeutic hypothermia is currently recommended in management of cardiac arrests with shockable rhythm. In mechanically ventilated patients who were resuscitated after out-of-hospital cardiac arrests, mild therapeutic hypothermia side effects are conductive for infectious complications and especially for ventilator-associated pneumonia (VAP).

Despite high incidence of VAP and other infectious complications, it is not currently recommended to use antibiotic prophylaxis on the responsible germs. Yet VAP incidence could be decreased if an antibiotic therapy was systematically given to patient treated with mild therapeutic hypothermia after a cardiac arrest. Several retrospective studies showed less infectious complications but also decreased morbidity and mortality related to these complications when antibiotic therapy was given early to patients treated with therapeutic hypothermia after cardiac arrest.

DETAILED DESCRIPTION:
Multicenter add-on randomized controlled double-blind trial assessing the efficacy of preventive antibiotics amoxicillin-clavulanic acid vs placebo to prevent occurrence of early VAP after out-of-hospital cardiac arrest receiving mild therapeutic hypothermia, in addition to usual VAP prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old, intubated and mechanically ventilated after out-of-hospital resuscitated cardiac arrest secondary to shockable rhythm
* Hospitalized in an ICU
* Mild therapeutic hypothermia procedure (32° to 35°C) scheduled (24 to 36 hours)
* Delay from ROSC to randomisation < 6 hours
* Consent from family members or emergency consent

Exclusion Criteria:

* Pregnancy
* Out-of-hospital cardiac arrest secondary to non shockable rhythm and In-hospital cardiac arrest
* Need for cardiac support by cardiopulmonary bypass
* Ongoing antibiotic therapy or during the week before
* Ongoing or concomitant pneumonia
* Known chronic colonization with MRB
* Hypersensitivity to the active substances, to any of the penicillins or to any of the excipients.
* History of a severe immediate hypersensitivity reaction (e.g. anaphylaxis) to another beta-lactam agent (e.g. a cephalosporin, carbapenem or monobactam).
* History of jaundice/hepatic impairment due to amoxicillin/clavulanic acid, according to the latest version of the SmPC.
* Previous lung disease
* Predictable decision of early care limitation
* Patient under guardianship or curatorship
* Moribund patient
* Participation to another trial within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Incidence reduction of early VAP | 7 days
  Incidence reduction of early VAP with short term amoxicillin-clavulanic acid in patients treated with hypothermia after out-of-hospital cardiac arrest

SECONDARY OUTCOMES:
Mortality | 28 days
  Mortality
Early nosocomial infectious complications | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FRANCOIS, MD, Principal Investigator — Limoges UH
Locations (16):
- France (16):
  - CH Angouleme - Service de Réanimation, Angoulême, Saint Michel
  - CH Argenteuil - Service de Réanimation, Argenteuil
  - CH Brive La Gaillarde - Service de Réanimation, Brive-la-Gaillarde
  - CHU Dijon - Serve de Réanimation, Dijon
  - AP-HP - Hôpital pointcaré - Service de Réanimation, Garches
  - CH du MANS, Le Mans
  - CHU de Limoges - Service de réanimation polyvalente, Limoges
  - CHU Nantes - Service de réanimation, Nantes
  - CHU Orléans - service de Réanimation, Orléans
  - AP-HP - Hôpital Lariboisière - Service de Réanimation, Paris
  - AP-HP - Hôpital Cochin - Service de Réanimation, Paris
  - AP-HP - Hôpital Européen Georges Pompidou - Service de Réanimation, Paris
  - CH Périgueux, Périgueux
  - CHU Strasbourg - service de Réanimation, Strasbourg
  - CHU Tours - Service de Réanimation, Tours
  - CH Versailles - service de Réanimation, Versailles

REFERENCES:
- [Result] Francois B, Cariou A, Clere-Jehl R, Dequin PF, Renon-Carron F, Daix T, Guitton C, Deye N, Legriel S, Plantefeve G, Quenot JP, Desachy A, Kamel T, Bedon-Carte S, Diehl JL, Chudeau N, Karam E, Durand-Zaleski I, Giraudeau B, Vignon P, Le Gouge A; CRICS-TRIGGERSEP Network and the ANTHARTIC Study Group. Prevention of Early Ventilator-Associated Pneumonia after Cardiac Arrest. N Engl J Med. 2019 Nov 7;381(19):1831-1842. doi: 10.1056/NEJMoa1812379. PMID 31693806